CLINICAL TRIAL: NCT04397081
Title: Comparison of Human Papilloma Virus Results in Women With and Without Atopic Disease
Brief Title: Atopic Diseases & Human Papilloma Virus
Status: Completed | Type: Observational
Sponsor: Adana Numune Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gulsum Uysal, Associate Professor in Obstetrics and Gynecology Department, Adana Numune Training and Research Hospital
Other Study IDs: 494/2019
Record Dates: First submitted 2020-05-17; First posted 2020-05-21 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Human Papilloma Virus; Atopic Asthma; Atopic Disorders
Keywords: Human papilloma virus,; screening test,; atopic diseases,; asthma,; rhinitis,; urticaria
MeSH Terms: conditions — Asthma; Rhinitis; Urticaria

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Control group was defined as healthy patients between the ages of 30-65 without allergic complaints.Patients' height, weight, demographic features (age, marital status, income level), obstetric histories (gravida, parity, mode of delivery), contraception methods and smoking status were noted.
  Interventions: Other: HPV test results
- Study group: Study group was defined as patients between the ages of 30-65 with allergic complaints complaints (sneezing, itching,runy nose, respiratory distress) were diagnosed "atopic disease" (allergic asthma, allergic rhinitis, allergic conjunctivitis, chronic urticaria and atopic dermatitis) by same clinician in Immunology and Allergy Department. Patients' height, weight, demographic features (age, marital status, income level), obstetric histories (gravida, parity, mode of delivery), contraception methods and smoking status were noted.
  Subgroup atopic disease diagnoses, duration of illness, treatments regimes and treatment time of the patients in the study group were also questioned and recorded.
  Interventions: Other: HPV test results

INTERVENTIONS:
Other: HPV test results — The human papillomavirus (HPV) test detects the presence of the human papillomavirus, a virus that can lead to the development of genital warts, abnormal cervical cells or cervical cancer. The procedure includes taking samples of your cervical cells using a soft brush and a flat scraping device called a spatula. This doesn't hurt, and you may not even feel the sample being taken.

SUMMARY:
Cervical cancer is an important health problem in women. Human papillomavirus (HPV) is considered the primary etiological agent of cervical cancer worldwide. Cervical cancer screening methods are proved one of the few screening methods that are thought to decrease invasive cancer incidence and mortality. In our country, HPV screening is carried out free of charge by public health to women between the ages of 30-65 aim is to compare HPV screening results between women diagnosed with atopic disease and healthy women without a history of atopy.If HPV is detected more frequently in patients with atopy, it may be recommended to follow more closely in vaccination and screening programs. Therefore, our study was designed to evaluate whether HPV positivity is common in atopic women.

DETAILED DESCRIPTION:
Patients between the ages of 30-65 with allergic complaints (sneezing, itching,runy nose, respiratory distress) were diagnosed "atopic disease" (allergic asthma, allergic rhinitis, allergic conjunctivitis, chronic urticaria and atopic dermatitis) by same clinician in Immunology and Allergy Department. Women aged between 30-65 years are scanned free of charge (HPV and smears) by the Public Health Institution in our country. The HPV results of the screened patients were noted retrospectively through the result reports of the patients, and those who were not screened were directed to Gynecology Department and HPV results were followed. Healthy women without allergic complaints applied for routine gynecologic examination occurred control group. Similarly, the HPV results of the control group were recorded.

Pregnant women, women who receive immunosuppressive therapy (including chemotherapy and chronic corticosteroid therapy), HIV positive women, women with cancer and performed hysterectomy were excluded. Patients' height, weight, demographic features (age, marital status, income level), obstetric histories (gravida, parity, mode of delivery), contraception methods and smoking status were noted.

Subgroup atopic disease diagnoses, duration of illness, treatments regimes and treatment time of the patients in the study group were also questioned and recorded. Leukotriene receptor antagonists and histamine receptor antagonists were the main treatments for study group and all therapies were designed by the same clinician. Routine allergic skin tests were performed to all atopic patients during diagnosis.

Statistical analyses

Statistical Package for Social Sciences (SPSS) for Windows, version 18.0 (SPSS Inc., USA) was used to compare the clinical features of groups. Normality of data distribution was tested with Kolmogorov-Smirnov test. Data was shown as means ± standart deviation (SD) for continuous variables and the independent t test was used to assess the differences in variables between groups. Kruskal-Wallis, Mann-Whitney U-test and Bonferroni correction were used for values with non-normal distribution. P Values below 0.05 (p<0.05) was accepted as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 30-65 with allergic complaints (sneezing, itching,runy nose, respiratory distress) diagnosed "atopic disease" (allergic asthma, allergic rhinitis, allergic conjunctivitis, chronic urticaria and atopic dermatitis) by same clinician in Immunology and Allergy Department.
* Patients between the ages of 30-65 without allergic complaints

Exclusion Criteria:

* Pregnant women
* women who receive immunosuppressive therapy (including chemotherapy and chronic corticosteroid therapy)
* HIV positive women
* women with cancer
* women performed hysterectomy

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 30-65 with allergic complaints (sneezing, itching,runy nose, respiratory distress) were diagnosed "atopic disease" (allergic asthma, allergic rhinitis, allergic conjunctivitis, chronic urticaria and atopic dermatitis) by same clinician in Immunology and Allergy Department. Healthy women without allergic complaints applied for routine gynecologic examination occurred control group.
Sampling Method: Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
to compare HPV screening results between women diagnosed with atopic disease and healthy women without a history of atopy. | 6 months
  comparing HPV test results between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Gulsum Uysal, Principal Investigator — Adana City Education and Research Hospital
Locations (1):
- Adana City Education and Research Hospital, Adana, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No